CLINICAL TRIAL: NCT06070324
Title: Effect of Suture Material on Postoperative Nipple Areolar Complex Widening: A Randomized Controlled Trial
Brief Title: Effect of Suture Material on Postoperative Nipple Areolar Complex Widening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Tanya DeLyzer, Co-Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123476
Record Dates: First submitted 2023-09-18; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Gynecomastia; Transgenderism; Breast Asymmetry
MeSH Terms: conditions — Breast Neoplasms; Gynecomastia; Transsexualism; Anisomastia | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: All patients will receive the surgical treatment they consented for, the only difference among them being the type of suture material used to close their perioareolar incisions (3 different types are investigated in this study).
Who Masked: Participant
Masking Description: The type of suture used to close the periareolar incision will be determined by drawing the name of the suture from a random, sealed envelope at the start of the procedure in the operating room. The patient will not be informed of the suture type and they are unable to see the suture type due to postoperative dressings being placed overtop, until they see the surgeon at their 2-week followup appointment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Prolene (Active Comparator): This group of patients will have their periareolar incisions closed with 4-0 Prolene sutures which are non-absorbable (require removal) and require knot-tying.
  Interventions: Procedure: Breast surgery; Device: Suturing of surgical incision
- Monocryl (Active Comparator): This group of patients will have their periareolar incisions closed with 4-0 Monocryl sutures which are absorbable (do not require removal) and require knot-tying.
  Interventions: Procedure: Breast surgery; Device: Suturing of surgical incision
- Stratafix (Active Comparator): This group of patients will have their periareolar incisions closed with 4-0 Stratafix sutures which are absorbable (do not require removal) and do not require knot-tying.
  Interventions: Procedure: Breast surgery; Device: Suturing of surgical incision

INTERVENTIONS:
Procedure: Breast surgery — Any surgery involving incisions made along the nipple areolar complex. These would include transgender mastectomy, cisgender female breast reduction/augmentation/reconstruction, and cisgender male gynecomastia correction.
Device: Suturing of surgical incision — The closing of a surgical incision by using sutures so appose and maintain apposition of two skin edges. Suturing may or may not require knot-tying depending on the material of suture used.

SUMMARY:
This will be a single-blinded study where participants are blinded to the suture type but the surgeon will draw a random, unmarked envelope containing the designated suture type at the start of the surgery. The patient population will be all patients undergoing breast surgery at the London Health Sciences Center (LHSC) - ie. University Hospital, Victoria Hospital and the Nazem Kadri Surgical Center, and St. Joseph's Hospital. Three (3) main procedure groups will be transgender gender-affirming top surgery, cisgender female breast reduction or augmentation (including healthy and cancer patients; subgroup analysis will be performed), and cisgender male gynecomastia surgery. The goal is n=180 patients, n=60 per type of suture with n=20 per type of procedure (totaling n=60 per type of procedure).

NAC width for each breast will be measured intraoperatively, at 2 weeks postop, 6 weeks postop, 3 months postop, and 6 months postop. These measurements will be deidentified and logged into a secure data entry form. Information on whether a secondary outcome occurred (ie. infection, dehiscence, revision and nipple necrosis) will be logged in this form as well.

Because the sutures will be kept non-visible under dressings until the clinical followup appointment 2 weeks postop, the patient will remain blinded as to the type of suture used on their NAC(s). At this point, absorbable sutures will have been largely dissolved and non-absorbable sutures will be removed.

DETAILED DESCRIPTION:
This will be a single-blinded study where the participants will be blinded to the type of suture. The patient population will be all patients undergoing breast surgery at the London Health Sciences Center (LHSC) - ie. University Hospital, Victoria Hospital and the Nazem Kadri Surgical Center - and St. Joseph's Hospital falling into one of 3 categories: transmasculine gender affirming top surgery, cisgender female elective or oncologic breast surgery (mastopexy, breast reduction, breast augmentation, or nipple-sparing mastectomy), and cisgender male gynecomastia correction.

Three sutures will be used: 4-0 Prolene, 4-0 Monocryl and 4-0 Stratafix. We will aim for n=180 participants, n=60 per type of suture, and n=60 per surgical category. This way, each suture type can be equally distributed among each surgical category. This means n=20 of each suture type will be used in n=20 of each surgery type. For example, n=20 top surgery patients will receive Prolene sutures, n=20 receive Monocryl, and n=20 receive Stratafix. All patients will be consented in the preop area on the day of their surgery by a member of the research team.

The primary outcomes will be NAC diameter or "width" intraoperatively immediately after closing compared to NAC width 2 weeks, 6 weeks, 3 months, and 6 months postoperatively. The horizontal and vertical widths will be measured at each time. Measurements are done with a ruler and recorded in centimeters. Prolene sutures will be removed at the 6-week postop visit as per current clinical practice. Absorbable will not be removed because they are absorbable.

Statistical regression will be used to determine whether a certain type(s) of suture is optimal for minimizing NAC widening after surgery. Subgroup analyses will also be conducted to determine any confounding factors from heterogeneity in patient factors within each group. Secondary outcomes will be rates of infection, tip loss, nipple necrosis and dehiscence, and whether certain types of sutures increase these adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any individual undergoing breast surgery of any kind using a periareolar approach including breast reconstruction, mastopexy, mammoplasty gender affirming surgery, mastectomy, or gynecomastia surgery
* Patients undergoing breast surgery at the London Health Sciences Center (LHSC) or St Joseph's Hospital (SJH)
* Participants over the age of 18
* Any BMI
* Any gender
* Patients who are willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Patient does not or cannot consent for enrollment in this study (includes inability to understand the provided information due to illiteracy or unproficiency in English)
* Patient is under the age of 18
* Patients with a known allergy to any type of suture material used in the study.
* For cancer patients who received radiotherapy, the irradiated breast will not be included in the study (the non-irradiated breast remains eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in nipple areolar complex diameter | 1 year
  Postoperative change in diameter of the nipple areolar complex as an adverse outcome

SECONDARY OUTCOMES:
Percentage of partial and nipple necrosis | 1 year
  Death of nipple tissue as an adverse outcome following surgery
Number of participants experiencing nipple tip loss | 1 year
  Loss of projection of the nipple tip due to effacement as an adverse outcome following surgery
Number of participants who contract a postoperative infection | 1 month
  Colonization of the surgical area by bacteria leading to immune response
Number of nipples that underwent incision dehiscence | 6 months
  Separation of the apposed skin edges along the surgical incision

IPD SHARING:
Plan to Share IPD: No